CLINICAL TRIAL: NCT03132233
Title: Safety, Tolerability and Efficacy of Exogenous Ketone Bodies for Preventive Treatment of Migraine: A Randomised, Placebo-controlled, Double-blind Study
Brief Title: Energy for the Brain
Acronym: MigraKet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: MigraKet
Record Dates: First submitted 2017-04-11; First posted 2017-04-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Migraine; Episodic Migraine
Keywords: Migraine; Prevention; Prophylaxis; Ketone bodies; Beta-hydroxybutyrate; Double-blind; Randomised; Placebo controlled; Mitochondrial functioning; Energy metabolism; Intervention; Dietary Supplement
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Active Comparator): Receives the investigational medicine product (IMP; Beta-hydroxybutyrate calcium and magnesium salt).
  Interventions: Dietary Supplement: Beta-hydroxybutyrate calcium and magnesium salt
- Placebo (Placebo Comparator): Receives a matched placebo powder to the IMP.
  Interventions: Other: placebo powder

INTERVENTIONS:
Dietary Supplement: Beta-hydroxybutyrate calcium and magnesium salt — Exogenous ketone body in mineral salt form.
  Arms: Verum
Other: placebo powder — matched placebo powder to the IMP.
  Arms: Placebo

SUMMARY:
Approx. one billion people are suffering from migraine worldwide and yet, therapeutic options are still very limited. Research suggests that changes in energy metabolism could be part of migraine pathophysiology. Ketone bodies (KB) are endogenous alternative energy substrates. Our clinical trial assesses the efficacy and safety of KB supplements in 60-90 adult migraineurs (5-14 migraine days / months) at the University Hospital Basel. The total duration of the trial is approx. 6 months, consisting of 4 weeks baseline, 12 weeks intervention with KB powder or matched placebo and 8 weeks follow-up. The primary endpoint is the change in migraine days at the end of intervention compared to baseline. Additionally, changes in gene expression, fat-, and glucose metabolism, inflammatory markers and quality of life will be examined.

DETAILED DESCRIPTION:
Migraine is a complex, common and debilitating neurological disorder. It affects approximately 17% of women and 8% of men in Europe and yet, its primary pathogenic mechanisms are still largely unknown. Various lines of research suggest that brain energy metabolism abnormalities are likely to be part of migraine pathophysiology. Specifically, there is some evidence for reversible abnormalities in mitochondrial functioning in migraine. For example, treatment with riboflavin and coenzyme Q10 has been shown to have migraine protective effects, probably via a positive effect on energy metabolism. Lactic and pyruvic acid, markers of mitochondrial (mt) disease, have been found to be increased in migraineurs; 31P-magnetic resonance spectroscopy (MRS) patterns seen in migraine are consistent with what is seen in mitochondrial disorders; cytochrome oxidase (COX)-negative fibres typical of mt diseases have also been seen in some patients with migraine. A break-down of the resting membrane potential due to lack of adenosine triphosphate (ATP) could explain cortical abnormalities in excitability, which have been reported in migraine. Despite causing a huge amount of suffering and a substantial amount of costs for society current migraine treatment options are limited. None of the prophylactic agents licensed to date are migraine-specific and most are associated with significant- sometimes intolerable- side-effects. Furthermore, their migraine-preventive properties are moderate at most. Hence, there is a need for developing alternative anti-migraine therapies. Several case studies and a first proof of concept study have demonstrated a reduction in migraine attack frequency, severity and use of acute anti-migraine medication during ketosis - with effects sizes ranging from total absence of attacks to a reduction to 1/5th of the run-in period. In addition, preliminary evidence suggests that the migraine-protective effect may outlast the duration of ketosis. This might be a result of longer-lasting gene-expression changes. However, a strict ketogenic diet (KD) is unlikely to provide a feasible long-term solution for episodic migraine patients, because it is difficult to implement in an ambulatory setting and patient adherence may be limited. An alternative means to induce a state of mild to medium nutritional ketosis (0.4-1 mmol/l), irrespective of blood glucose levels, is the dietary supplementation with ketogenic substances, such as beta-hydroxybutyrate (bHB) salts (and unpublished observations). This approach could be easily implemented with intake of a ketogenic powder dissolved in water (consisting of a calcium-magnesium-bHB salt) three times a day (with or after a meal). This nutritional intervention seems much more feasible than a KD in larger patient populations and avoids the complications of a very restricted high-fat diet.

ELIGIBILITY:
Inclusion Criteria:

* Has been previously diagnosed with migraine (with or without aura) in accordance with the ICHD-3 Beta Classification criteria.
* Experience between 5 and 14 migraine days per month (over the last 4 months).
* Has age of onset of migraine less than 50 years old.
* Agrees to refrain from initiating or changing the type, dosage or frequency of any prophylactic medications (exclusive of medications taken for acute relief of migraine symptoms) as well as dietary supplements (such as Q10, riboflavin etc) against migraine and for indications other than migraine that in the opinion of the clinician may interfere with the study objectives (e.g. antidepressant, anticonvulsants, beta blockers, etc.) for the duration of the study.
* Has not changed type, dosage or frequency of any prophylactic medications (exclusive of medications taken for acute relief of migraine symptoms) as well as dietary supplements (such as Q10, riboflavin etc) against migraine and for indications other than migraine that in the opinion of the clinician may interfere with the study objectives (e.g. antidepressant, anticonvulsants, beta blockers, etc.) for at least 3 months prior to study onset.
* Refrains to make any drastic changes to the diet for the duration of the study, including periods of fasting.
* Agrees to use the study intervention as intended, follow all of the requirements of the study including follow-up visit requirements, record required study data in the subject dairy and other self-assessment questionnaires and is okay with drawing blood samples.
* Is able to provide written Informed Consent.

Exclusion Criteria:

* Has a concomitant medical condition that will require oral or injectable steroids during the study.
* Has a history of any significant neurological, psychiatric or other medical condition that in the opinion of the investigator may confound the study assessments, liver and kidney diseases in particular.
* Is currently treated for a thyroid disease or has a history thereof.
* Has a cardiovascular disease (hypertension in particular) or a history thereof.
* Has a known history of suspected secondary headache.
* Currently takes simple analgesics or non-steroidal anti-inflammatory drugs (NSAIDs) greater then 14 days per month or triptans greater than 10 days per month for headaches or other body pain.
* Currently takes prescription opioids.
* Has previous diagnosis of medication overuse headache (MoH) , which has reverted to episodic migraine within the last 6 months.
* Meets the ICHD-3 Beta Classification criteria for chronic migraine (> 15 headache days per month).
* Has failed an adequate trial (two months or greater) of at least 3 classes of a drug therapy for the prophylaxis of migraine .
* Has had surgery for migraine prevention.
* Has received Botox injections within the last 6 months.
* Is pregnant or thinking of becoming pregnant during the study period, or of childbearing years and is unwilling to use and accepted form of birth control.
* Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
* Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self- assessments is compromised (e.g. homeless, developmentally disabled and prisoner).
* Is thinking to start, change or stop a hormone-based contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Number of migraine days | Last 4 weeks of intervention compared to baseline 4 weeks.
  Mean change from baseline in number of migraine days (meeting International Classification of Headache Disorders (ICHD)-3 criteria) during the last month of intervention in treatment group compared to placebo.

SECONDARY OUTCOMES:
Number of headache days | Last 4 weeks of intervention compared to baseline 4 weeks.
  Mean change from baseline in number of headache days of any severity (meeting ICHD-3 criteria) during the last month of intervention in treatment group compared to placebo.
Acute migraine medication | Last 4 weeks of intervention compared to baseline 4 weeks.
  Mean change from baseline in consumption of acute migraine medication (analgesics or triptans) measured in days with acute headache medication use during the last month of the intervention.
Migraine intensity | Last 4 weeks of intervention compared to baseline 4 weeks.
  Mean change from baseline in migraine intensity (measured with a numerical rating scale from 1-10) during the last of month of the intervention period.
Migraine Disability Assessment (MIDAS) | Last 4 weeks of intervention compared to baseline 4 weeks.
  Score in Migraine Disability Assessment (MIDAS; end of baseline versus end of intervention).
Headache Impact Test (HIT) | Last 4 weeks of intervention compared to baseline 4 weeks.
  Score in Headache Impact Test (HIT-6; end of baseline versus end of intervention).

OTHER OUTCOMES:
Exploratory biomarker assessments | Last 4 weeks of intervention compared to baseline 4 weeks.
  Serum concentration changes from baseline of oxidative and nitrosative stress markers (malondialdehyde (MDA), carbonylated proteins, nitrate, nitrite, nitrotyrosine), levels in cytokines, levels in lactate, glucose, insulin and markers of thyroid function. Genetic profile (SNPs) of all patients involved in the study and correlation of the genetic markers with 1-5 using a linear regression model. Gene expression changes before and after diet using expression microarrays with a special focus on mitochondrial related genes (Citrate synthesis, Cytochrom C oxidase subunit 1, Succinate dehydrogenase subunit A). Correlation of gene expression changes with the genetic profile of the patients (eQTL analysis in combination with 1-5 as possible covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Fischer, MD, Principal Investigator — Professor and head doctor
Locations (1):
- University Children's Hospital (UKBB), Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Putananickal N, Gross EC, Orsini AL, Schmidt S, Hafner P, Gocheva V, Nagy S, Henzi BC, Rubino D, Schadelin S, Sandor P, Fischer D. Metabolic markers of short and long-term exogenous DL-beta-hydroxybutyrate supplementation in episodic migraine patients: an exploratory analysis of a randomized-controlled-trial. Front Pharmacol. 2023 May 4;14:1172483. doi: 10.3389/fphar.2023.1172483. eCollection 2023. PMID 37214431
- [Derived] Gross EC, Putananickal N, Orsini AL, Schoenen J, Fischer D, Soto-Mota A. Defining metabolic migraine with a distinct subgroup of patients with suboptimal inflammatory and metabolic markers. Sci Rep. 2023 Mar 7;13(1):3787. doi: 10.1038/s41598-023-28499-y. PMID 36882474
- [Derived] Putananickal N, Gross EC, Orsini AL, Schmidt S, Hafner P, Gocheva V, Nagy S, Henzi BC, Rubino D, Vogt DR, Cichon S, Sandor P, Fischer D. Efficacy and safety of exogenous beta-hydroxybutyrate for preventive treatment in episodic migraine: A single-centred, randomised, placebo-controlled, double-blind crossover trial. Cephalalgia. 2022 Apr;42(4-5):302-311. doi: 10.1177/03331024211043792. Epub 2021 Sep 20. PMID 34541914
- [Derived] Gross EC, Putananickal N, Orsini AL, Vogt DR, Sandor PS, Schoenen J, Fischer D. Mitochondrial function and oxidative stress markers in higher-frequency episodic migraine. Sci Rep. 2021 Feb 25;11(1):4543. doi: 10.1038/s41598-021-84102-2. PMID 33633187
- [Derived] Gross E, Putananickal N, Orsini AL, Schmidt S, Vogt DR, Cichon S, Sandor P, Fischer D. Efficacy and safety of exogenous ketone bodies for preventive treatment of migraine: A study protocol for a single-centred, randomised, placebo-controlled, double-blind crossover trial. Trials. 2019 Jan 17;20(1):61. doi: 10.1186/s13063-018-3120-7. PMID 30654835
- See also: Study Information Video — https://www.youtube.com/watch?v=2YzNjIXk_eY